CLINICAL TRIAL: NCT01889069
Title: A Single Arm, Multicentre, Phase IIIB Study to Evaluate Safety, Efficacy and Pharmacokinetic (PK) of Subcutaneous (SC) Rituximab Administered During Induction Phase or Maintenance in Previously Untreated Patients With CD20+ Diffuse Large B Cell Lymphoma (DLBCL) or Follicular Lymphoma (FL)
Brief Title: A Study to Evaluate Safety, Efficacy and Pharmacokinetics of Rituximab (MabThera/Rituxan) in Participants With Diffuse Large B Cell Lymphoma (DLBCL) or Follicular Lymphoma (FL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28881; 2013-000647-12 (EudraCT Number)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisone; Bendamustine Hydrochloride

ARMS (1):
- Rituximab (Experimental): Participants will receive at least 4 doses of rituximab 1400 mg SC once a month during the Induction period, and at least 6 doses of rituximab 1400 mg SC once every two months during the Maintenance period, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); or bendamustine as per standard local practice.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisone; Drug: Bendamustine

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered at a dose of 1400 mg SC once a month for at least 4 doses during the Induction period, and at a dose of 1400 mg SC once every two months for at least 6 doses during the Maintenance period.
  Other Names: MabThera; Rituxan
Drug: Cyclophosphamide — Cyclophosphamide will be administered as per standard local practice as a part of standard chemotherapy regimen.
Drug: Vincristine — Vincristine will be administered as per standard local practice as a part of standard chemotherapy regimen.
Drug: Doxorubicin — Doxorubicin will be administered as per standard local practice as a part of standard chemotherapy regimen.
Drug: Prednisone — Prednisone will be administered as per standard local practice as a part of standard chemotherapy regimen.
Drug: Bendamustine — Bendamustine will be administered as per standard local practice as a part of standard chemotherapy regimen.

SUMMARY:
This single arm, multicenter study will evaluate the safety, efficacy and pharmacokinetic (PK) of subcutaneous (SC) rituximab in previously untreated participants with cluster of differentiation 20 positive (CD20+) DLBCL or FL. In addition to standard chemotherapy, participants will receive at least 4 doses of rituximab 1400 mg SC once a month during the Induction period, and at least 6 doses of rituximab 1400 mg SC once every two months during the Maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, CD20+ DLBCL or CD20+ follicular non-Hodgkin's lymphoma (NHL) Grade 1, 2 or 3a, according to the World Health Organization (WHO) classification system
* Currently being treated with rituximab intravenously (IV) in the Induction or Maintenance period, having received at least one full dose of rituximab IV, defined as standard full dose of rituximab IV 375 milligrams per square-meter (mg/m^2) administered without interruption or early discontinuation (i.e. tolerability issues)
* Expectation and current ability for the participant to receive at least 4 additional cycles of treatment during the Induction period or 6 additional cycles of treatment during the Maintenance period (participants with follicular NHL)
* An International Prognostic Index (IPI) score of 1-4 or IPI score of 0 with bulky disease, defined as one lesion greater than or equal to (>=) 7.5 centimeters (cm), or Follicular Lymphoma International Prognostic Index (FLIPI) (low, intermediate or high risk) assessed before the first rituximab IV administration in Induction period
* At least one bi-dimensionally measurable lesion defined as >=1.5 cm in its largest dimension on computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (<=) 3

Exclusion Criteria:

* Transformed lymphoma or FL IIIB
* Primary central nervous system lymphoma, histologic evidence of transformation to a Burkitt lymphoma, primary effusion lymphoma, primary mediastinal DLBCL, DLBCL of the testis, or primary cutaneous DLBCL
* History of other malignancy
* Ongoing corticosteroid use greater than (>) 30 milligrams per day (mg/day) of prednisone or equivalent
* Inadequate renal, hematologic, or hepatic function
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindications to any of the individual components of standard chemotherapy
* Other serious underlying medical conditions, which, in the Investigator's judgement, could impair the ability of the participant to participate in the study
* Recent major surgery (within 4 weeks prior to dosing, other than for diagnosis)
* Active hepatitis B virus (HBV), active hepatitis C virus (HCV) infection, or human immunodeficiency virus (HIV) infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Italy (39):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Azienda ospedaliera oo rr di foggi; Hematology, Foggia, Apulia
  - Irccs Crob, Rionero in Vulture, Basilicate
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli; Unità Operativa di Ematologia, Reggio Calabria, Calabria
  - Azienda Ospedaliera S.G. Moscati; Divisione Ematologia, Avellino, Campania
  - Asl ce - p.o. Avers; Uoc ematologia, Aversa, Campania
  - A.O. San Sebastiano; U.O.C. Oncologia, Caserta, Campania
  - Seconda università degli studi di napoli; Medicina clinica e sperimentale magrassi - lanzara, Napoli, Campania
  - Osp. Santa Maria Goretti; Ematologia, Latina, Lazio
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Regina Elena National Cancer Institute; Hematology, Rome, Lazio
  - Az. Osp. S. Camillo Forlanini; Uo Ematologia E Trapianti Di Midollo Osseo, Rome, Lazio
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia; Dip Biot Cel e Ematol, Rome, Lazio
  - Azienda Ospedaliera S. Giovanni Addolorata; UOC Ematologia, Rome, Lazio
  - ASL Viterbo; Presidio Ospedaliero di Ronciglione; UOC Ematologia, Ronciglione, Lazio
  - Ospedale Valduce;U.O.S. Oncologia Ed Ematologia, Como, Lombardy
  - ASST DI CREMA; U O Oncologia Medica, Crema, Lombardy
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - Az. Osp. Carlo Poma; Divisione Di Oncologia Medica, Mantova, Lombardy
  - Osp. San Raffaele; Dip. Di Oncoematologia, Milan, Lombardy
  - Ist. Nazionale Per Lo Studio E Cura Dei Tumori; Div. Ematologia Trapianto Midollo Osseo Allogenico, Milan, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Università Cattolica Del Sacro Cuore S.S. Giovanni Paolo Ii; Uoc Di Onco-Ematologia, Campobasso, Molise
  - Ospedale Civile SS. Antonio E Biagio DI Alessandria; Ematologia, Alessandria, Piedmont
  - Univ. Piemonte Est Amedeo Avogadro; Div.Ematologia- Dip.Clinica Med.Sperim.& Ircad, Novara, Piedmont
  - Ospedale Roberto Binaghi; Centro trapianti di midollo osseo, Cagliari, Sardinia
  - Osp. San Francesco; Ematologia e CTMO, Nuoro, Sardinia
  - ARNAS Garibaldi; Ematologia, Catania, Sicily
  - Az. Osp. Papardo; Struttura Complessa Di Ematologia, Messina, Sicily
  - ARNAS-Ospedale Civico Maurizio Ascoli; Unità Operativa di Oncologia Medica, Palermo, Sicily
  - Azienda Uni Ria Policlinico P. Giaccone ; Divisione Di Ematologia E Trapianto, Palermo, Sicily
  - Ospedale Gen.Le Prov.Le 'C.G.Mazzoni'; Ematologia, Ascoli Piceno, The Marches
  - Ospedale di Civitanova Marche; Medicina Interna, Civitanova Marche, The Marches
  - Ospedale di Macerata; Medicina Generale, Macerata, The Marches
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
  - USL 4 di Prato - Nuovo Ospeale di Prato, Prato, Tuscany
  - A.O. Santa Maria Terni; S.C. Oncoematologia, Terni, Umbria
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 37 investigational centers in Italy.
Pre-assignment Details: Total overall participants enrolled in the study was 159, however for the subject disposition and baseline characteristics the enrolled was 158 as one participant discontinued the study prior to treatment.
Groups:
- Subcutaneous (SC) Rituximab: Participants will receive at least 4 doses of rituximab 1400 mg SC once a month during the Induction period, and at least 6 doses of rituximab 1400 mg SC once every two months during the Maintenance period, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); or bendamustine as per standard local practice.
Period: Overall Study
Arm/Group | Subcutaneous (SC) Rituximab
Started (All Enrolled Participants) | 158
Completed | 113
Not Completed | 45
Not completed — Death | 18
Not completed — Progression of Disease | 14
Not completed — Lost to Follow-up | 6
Not completed — Other | 4
Not completed — Consent Withdrawal | 3

BASELINE CHARACTERISTICS:
Population: ITT population included all enrolled participants. All analyses described have been performed by type of lymphoma (DLBCL/ FL) and overall. Total overall participants enrolled in the study was 159, however for the subject disposition and baseline characteristics the enrolled was 158 as one participant discontinued the study prior to treatment.
Groups:
- Diffuse Large B-Cell Lymphoma (DLBCL): Participants with DLBCL, who had received at least 4 doses of rituximab 1400 mg SC once a month during the treatment phase, up to a maximum of 7 cycles, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); as per standard local practice.
- Follicular Lymphoma (FL): Participants with CD20+ non-Hodgkin's (FL), who had received at least 4 doses of rituximab 1400 mg SC once a month during the Induction period, and at least 6 doses of rituximab 1400 mg SC once every two months during the Maintenance period, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); or bendamustine as per standard local practice.
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Total
Number analyzed (Participants) | 72 | 86 | 158
Age, Continuous [Mean (Standard Deviation); unit: years]
  Intent-to-Treat Population | 59.7 (12.70) | 57.8 (9.92) | 58.7 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 44 | 72
  Male | 44 | 42 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 59 | 72 | 131
  Unknown or Not Reported | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Administration-Associated Reactions (AAR)
Description: AARs were defined as all adverse events (AEs) occurring within 24 hours of rituximab administration and which were considered related to study drug. AARs included infusion/injection-related reactions (IIRRs), injection-site reactions, administration site conditions and all symptoms thereof. Grading was completed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: Baseline up to 54 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Groups:
- Diffuse Large B-Cell Lymphoma (DLBCL): Participants with DLBCL, who had received at least 4 doses of rituximab 1400 mg SC once a month during the treatment phase, up to a maxium of 7 cycles, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); as per standard local practice.
- Subcutaneous (SC) Rituximab: Participants with CD20+ diffuse large B-cell lymphoma (DLBCL) or non-Hodgkin's follicular lymphoma (FL), who received at least 4 doses of rituximab 1400 mg SC once a month during the Induction period, and at least 6 doses of rituximab 1400 mg SC once every two months during the Maintenance period, in addition to standard chemotherapy. Standard chemotherapy regimen included cyclophosphamide, vincristine, doxorubicin and prednisone (CHOP); or cyclophosphamide, vincristine and prednisone (CVP); or bendamustine as per standard local practice.
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants
  At least One AAR | 4.2 | 8.1 | 6.3
  At Least One AAR Grade ≥3 | 0 | 0 | 0
  Cutaneous and Soft Tissue AARs (Localized) | 1.4 | 8.1 | 5.1
  Cutaneous and Soft Tissue AARs (Non-Localized) | 2.8 | 0 | 1.3

2. Secondary Outcome: Percentage of Participants With At Least One Grade ≥ 3 Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with the treatment. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study were also considered as adverse events. Grading was completed according to the CTCAE, version 4.0.
Time Frame: Baseline up to 54 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 51.4 | 43.0 | 46.8

3. Secondary Outcome: Percentage of Participants With At Least One Grade ≥ 3 Infusion/ Injection Related Reactions (IIRRs)
Description: Grading of IIRRs was completed according to the CTCAE, version 4.0.
Time Frame: Baseline up to 54 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With At Least One Treatment-Emergent Serious Adverse Events
Description: SAE was defined as any experience that suggested a significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/ birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: Baseline up to 54 months
Population: Safety Population included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 36.1 | 26.7 | 31.0

5. Secondary Outcome: Percentage of Participants With Event-Free Survival (EFS) According to IWG Response Criteria
Description: EFS was defined as the time from first dose of rituximab to first occurrence of progression or relapse, according to the International Working Group (IWG) response criteria or other country standards, or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurred first.
Time Frame: Day 1 up to first occurrence of progression or relapse, or initiation of a non-protocol-specified anti-lymphoma therapy or death, whichever occurs first (up to maximum 54 months)
Population: ITT population included all enrolled participants who received at least one dose of the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 29.2 | 22.1 | 25.3

6. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) According to IWG Response Criteria
Description: PFS was defined as the time from first dose of rituximab to the first occurrence of disease progression or relapse, according to the International Working Group (IWG) response criteria or other country standards, or death from any cause, whichever occurred first.
Time Frame: Day 1 up to first occurrence of progression or relapse, or death, whichever occurs first (up to maximum 54 months)
Population: ITT population included all enrolled participants who received at least one dose of the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 29.2 | 22.1 | 25.3

7. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS was defined as the time from first dose of rituximab to death from any cause.
Time Frame: Day 1 until death (up to maximum 54 months)
Population: ITT population included all enrolled participants who received at least one dose of the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 19.4 | 4.7 | 11.4

8. Secondary Outcome: Percentage of Participants With Disease-Free Survival (DFS) According to IWG Response Criteria
Description: DFS assessed in participants achieving complete response (CR) including complete response unconfirmed (Cru) and was defined as the period from 4 to 8 weeks after end of Induction period up to relapse or death from any cause, whichever occured first.
Time Frame: From 4 to 8 weeks after end of Induction period up to relapse or death from any cause, whichever occurs first (up to maximum 54 months) (end of Induction period = up to 8 months)
Population: ITT population included all enrolled participants who received at least one dose of the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 21.7 | 25.6 | 23.5

9. Secondary Outcome: Percentage of Participants With Complete Response (CR) According to IWG Response Criteria
Description: Complete response required: 1) the complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities, 2) all lymph nodes and nodal masses had regressed to normal size, 3) the spleen, if considered to be enlarged before therapy on the basis of a CT scan, must have regressed in size and not be palpable on physical examination and 4) if the bone marrow was involved by lymphoma before treatment, the infiltrate was cleared on repeat bone marrow aspirate and biopsy of the same site. CR/unconfirmed (CRu) included those patients who fulfilled criteria 1 and 3 above as well as 1) a residual lymph node mass greater than 1.5 cm in greatest transverse diameter that regressed by more than 75% in the SPD and 2) indeterminate bone marrow. Response was assessed according to the IWG response criteria.
Time Frame: At 4 to 8 weeks after end of Induction period (end of Induction period = up to 8 months)
Population: ITT population included all enrolled participants who received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL) | Subcutaneous (SC) Rituximab
Number analyzed (Participants) | 72 | 86 | 158
Percentage of Participants | 65.2 [52.4 to 76.5] | 67.9 [53.7 to 80.1] | 66.4 [57.2 to 74.8]

10. Secondary Outcome: FL: Plasma Trough Concentrations of Rituximab
Description: FL participants could be enrolled during induction or maintenance phase and they should have received at least 1 infusion of rituximab and must have been able to receive at least 4 cycles of rituximab SC if enrolled during induction or 4 cycles of rituximab SC if enrolled during maintenance. Pharmacokinetic (PK) data only collected for participants enrolled during Induction. During the induction phase each Cycle is 21 days.
Time Frame: Induction collection: Cycle 2 Predose, Cycle 3 Predose, Cycle 4 Predose, Cycle 5 Predose, Baseline Predose, and Cycle 8 Predose on Day 1
Population: The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Follicular Lymphoma (FL)
Number analyzed (Participants) | 31
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 10
  Cycle 2 Predose | 55.49 (64.275)
  Cycle 3 Predose: number analyzed (Participants) | 6
  Cycle 3 Predose | 119.50 (139.606)
  Cycle 4 Predose: number analyzed (Participants) | 4
  Cycle 4 Predose | 157.25 (132.583)
  Cycle 5 Predose: number analyzed (Participants) | 1
  Cycle 5 Predose | 7.60 (NA) — Standard deviation could not be calculated from data for a single participant.
  Baseline: number analyzed (Participants) | 21
  Baseline | 90.88 (107.089)
  Cycle 8 Predose: number analyzed (Participants) | 23
  Cycle 8 Predose | 201.56 (372.609)

11. Secondary Outcome: FL: Overall Geometric Least Square (LS) Mean Plasma Trough Concentrations of Rituximab
Description: FL participants could be enrolled during induction or maintenance phase and they should have received at least 1 infusion of rituximab and must have been able to receive at least 4 cycles of rituximab SC if enrolled during induction or 4 cycles of rituximab SC if enrolled during maintenance. PK data only collected for participants enrolled during Induction. During the induction phase each Cycle is 21 days.
Time Frame: as for outcome 10
Population: The overall geometric LS mean plasma trough concentrations of rituximab in participants with FL in the pharmacokinetic (PK) population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: micrograms per millilitre (ug/mL)
Arm/Group | Follicular Lymphoma (FL)
Number analyzed (Participants) | 31
micrograms per millilitre (ug/mL) | 61.01 [42.49 to 87.61]

12. Secondary Outcome: FL: Plasma Trough Concentrations of Rituximab in Participants With Complete Response/Complete Response Unconfirmed (CR/CRu)
Description: as for outcome 11
Time Frame: as for outcome 10
Population: FL participants with Complete Response/Complete Response Unconfirmed (CR/CRu). The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Follicular Lymphoma (FL)
Number analyzed (Participants) | 20
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 8
  Cycle 2 Predose | 48.86 (57.640)
  Cycle 3 Predose: number analyzed (Participants) | 3
  Cycle 3 Predose | 156.33 (193.753)
  Cycle 4 Predose: number analyzed (Participants) | 3
  Cycle 4 Predose | 200.33 (123.411)
  Cycle 5 Predose: number analyzed (Participants) | 1
  Cycle 5 Predose | 7.60 (NA) — Standard deviation could not be calculated from data for a single participant.
  Baseline: number analyzed (Participants) | 15
  Baseline | 97.90 (118.897)
  Cycle 8 Predose: number analyzed (Participants) | 12
  Cycle 8 Predose | 284.08 (504.113)

13. Secondary Outcome: DLBCL: Plasma Concentrations of Rituximab
Description: DLBCL participants received at least 1 infusion of rituximab and must have been able to receive at least 4 cycles of rituximab SC; therefore DLBCL participants could be enrolled at Cycle 2, Cycle 3, Cycle 4, or Cycle 5 and as a result the baseline PK sample could be collected at Cycle 2, Cycle 3, Cycle 4, or Cycle 5. Each Cycle is 21 days.
Time Frame: Cycle 2 Predose, Cycle 3 Predose, Cycle 4 Predose, Cycle 5 Predose, Baseline Predose, Cycle 7 Predose on Day 1, Cycle 7 Day 7, Cycle 7 Day 14, Cycle 8 Predose on Day 1
Population: The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 10
  Cycle 2 Predose | 42.53 (49.637)
  Cycle 3 Predose: number analyzed (Participants) | 9
  Cycle 3 Predose | 88.92 (92.790)
  Cycle 4 Predose: number analyzed (Participants) | 2
  Cycle 4 Predose | 110.50 (101.116)
  Cycle 5 Predose: number analyzed (Participants) | 5
  Cycle 5 Predose | 100.20 (44.483)
  Baseline: number analyzed (Participants) | 30
  Baseline | 92.92 (114.466)
  Cycle 7 Predose: number analyzed (Participants) | 26
  Cycle 7 Predose | 141.44 (122.314)
  Cycle 7 Day 7: number analyzed (Participants) | 20
  Cycle 7 Day 7 | 348.81 (490.785)
  Cycle 7 Day 14: number analyzed (Participants) | 5
  Cycle 7 Day 14 | 226.40 (136.729)
  Cycle 8 Predose: number analyzed (Participants) | 28
  Cycle 8 Predose | 117.61 (89.394)

14. Secondary Outcome: DLBCL: Plasma Trough Concentrations of Rituximab
Description: as for outcome 13
Time Frame: Cycle 2 Predose, Cycle 3 Predose, Cycle 4 Predose, Cycle 5 Predose, Baseline Predose, Cycle 7 Predose on Day 1, Cycle 7 Day 7, Cycle 7 Day 14, Cycle 8 pre-dose on Day 1
Population: The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 10
  Cycle 2 Predose | 42.53 (49.637)
  Cycle 3 Predose: number analyzed (Participants) | 9
  Cycle 3 Predose | 88.92 (92.790)
  Cycle 4 Predose: number analyzed (Participants) | 2
  Cycle 4 Predose | 110.50 (101.116)
  Cycle 5 Predose: number analyzed (Participants) | 5
  Cycle 5 Predose | 100.20 (44.483)
  Baseline: number analyzed (Participants) | 30
  Baseline | 92.92 (114.466)
  Cycle 7 Predose: number analyzed (Participants) | 26
  Cycle 7 Predose | 141.44 (122.314)
  Cycle 8 Predose: number analyzed (Participants) | 21
  Cycle 8 Predose | 117.61 (89.394)

15. Secondary Outcome: DLBCL: Area Under the Plasma Concentration-Time Curve (AUC) of Rituximab
Description: as for outcome 13
Time Frame: as for outcome 13
Population: PK evaluable population. AUC was not estimable for available PK concentrations in DLBCL participants.
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
mcg*hr/mL | NA (NA) — AUC was not estimable for available PK concentrations in DLBCL participants

16. Secondary Outcome: DLBCL: Maximum Plasma Concentration (Cmax) of Rituximab
Description: as for outcome 13
Time Frame: as for outcome 13
Population: PK evaluable population. Cmax was not estimable for available PK concentrations in DLBCL participants.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
micrograms per millilitre (ug/mL) | NA (NA) — Cmax was not estimable for available PK concentrations in DLBCL participants.

17. Secondary Outcome: DLBCL: Apparent Total Clearance (CL/F) of Rituximab
Description: as for outcome 13
Time Frame: as for outcome 13
Population: PK evaluable population. CL/F was not estimable for available PK concentrations in DLBCL participants.
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
liter per hour (L/h) | NA (NA) — CL/F was not estimable for available PK concentrations in DLBCL participants.

18. Secondary Outcome: DLBCL: Plasma Trough Concentrations of Rituximab in Participants With Complete Response/Complete Response Unconfirmed (CR/CRu)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: DLBCL participants with Complete Response/Complete Response Unconfirmed (CR/CRu). The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 28
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 7
  Cycle 2 Predose | 53.97 (56.169)
  Cycle 3 Predose: number analyzed (Participants) | 7
  Cycle 3 Predose | 101.79 (101.223)
  Cycle 4 Predose: number analyzed (Participants) | 2
  Cycle 4 Predose | 110.50 (101.116)
  Cycle 5 Predose: number analyzed (Participants) | 3
  Cycle 5 Predose | 121.67 (45.092)
  Baseline: number analyzed (Participants) | 23
  Baseline | 109.40 (125.603)
  Cycle 7 Predose: number analyzed (Participants) | 21
  Cycle 7 Predose | 157.93 (131.178)
  Cycle 8 Predose: number analyzed (Participants) | 21
  Cycle 8 Predose | 132.57 (95.447)

19. Secondary Outcome: DLBCL: Overall Geometric Least Square (LS) Mean Plasma Trough Concentrations of Rituximab
Description: as for outcome 13
Time Frame: as for outcome 13
Population: The overall geometric LS mean plasma trough concentrations of rituximab in participants with DLBCL in the PK population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: micrograms per millilitre (ug/mL)
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 36
micrograms per millilitre (ug/mL) | 70.50 [57.60 to 86.28]

20. Secondary Outcome: DLBCL: Plasma Concentrations During Different Scheduling of Rituximab SC R-CHOP-14 or R-CHOP-21
Description: Plasma concentrations of rituximab in participants with DLBCL by chemotherapy regimen cyclophosphamide, oncovine (vincristine), doxorubicin, prednisone/prednisolone given every 14 days (R-CHOP-14) or cyclophosphamide, oncovine (vincristine), doxorubicin, prednisone/prednisolone given every 21 days (R-CHOP-21) in the PK) population.DLBCL participants received at least 1 infusion of rituximab and must have been able to receive at least 4 cycles of rituximab SC; therefore DLBCL participants could be enrolled at Cycle 2, Cycle 3, Cycle 4, or Cycle 5 and as a result the baseline PK sample could be collected at Cycle 2, Cycle 3, Cycle 4, or Cycle 5. Each Cycle is 21 days.
Time Frame: as for outcome 13
Population: DLBCL: R-CHOP 21 or R-CHOP-14; The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Groups:
- Diffuse Large B-Cell Lymphoma (DLBCL) R-CHOP-14: Cyclophosphamide, oncovine (vincristine), doxorubicin, prednisone/prednisolone given every 14 days
- Diffuse Large B-Cell Lymphoma (DLBCL) R-CHOP-21: Cyclophosphamide, oncovine (vincristine), doxorubicin, prednisone/prednisolone given every 21 days
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) R-CHOP-14 | Diffuse Large B-Cell Lymphoma (DLBCL) R-CHOP-21
Number analyzed (Participants) | 4 | 31
micrograms per millilitre (ug/mL)
  Cycle 2 Predose: number analyzed (Participants) | 1 | 9
  Cycle 2 Predose | 170.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 28.37 (22.695)
  Cycle 3 Predose: number analyzed (Participants) | 0 | 9
  Cycle 3 Predose |  | 88.92 (92.790)
  Cycle 4 Predose: number analyzed (Participants) | 0 | 2
  Cycle 4 Predose |  | 110.50 (101.116)
  Cycle 5 Predose: number analyzed (Participants) | 1 | 4
  Cycle 5 Predose | 125.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 94.00 (48.806)
  Baseline: number analyzed (Participants) | 4 | 26
  Baseline | 214.25 (233.493) | 74.25 (77.064)
  Cycle 7 Predose: number analyzed (Participants) | 2 | 23
  Cycle 7 Predose | 93.50 (79.903) | 150.13 (126.221)
  Cycle 7 Day 7: number analyzed (Participants) | 2 | 17
  Cycle 7 Day 7 | 71.55 (26.092) | 398.76 (517.974)
  Cycle 7 Day 14: number analyzed (Participants) | 1 | 4
  Cycle 7 Day 14 | 42.00 (NA) — Standard deviation could not be calculated from data for a single participant. | 272.50 (103.722)
  Cycle 8 Predose: number analyzed (Participants) | 2 | 25
  Cycle 8 Predose | 78.50 (14.849) | 123.76 (92.606)

21. Secondary Outcome: Rituximab Administration Satisfaction Questionnaire (RASQ) Convenience and Satisfaction Domain Scores
Description: Patient-assessed satisfaction was evaluated using RASQ. Participants were asked questions regarding convenience and satisfaction for rituximab SC. Each domain is scored on a scale of 0 to 100, with higher scores indicative of more positive feelings toward therapy. The score for each domain was averaged among all participants. DLBCL participants could be enrolled at cycle 2, cycle 3, or cycle 4. FL participants could be enrolled during induction or maintenance phase and they should have received at least 1 infusion of rituximab and must be able to receive at least 4 cycles of rituximab SC if enrolled during induction or 4 cycles of rituximab SC if enrolled during maintenance. Each Cycle is 21 days for DLBCL. Each Cycle 21 days during the Induction phase and 2 months during Maintenance phase for FL.
Time Frame: DLBCL: Cycle (C) 2, C3, C4, C5, C6, End of C8; FL: Induction: C3, C4, C5, C6, C8, Maintenance: C2, C3, C4, C5, C6, C7, C8, C10, C12, End of treatment (4-8 weeks after last dose)
Population: Safety population included all enrolled patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL)
Number analyzed (Participants) | 72 | 86
Units on a Scale
  Convenience domain Cycle 3 Induction: number analyzed (Participants) | 0 | 27
  Convenience domain Cycle 3 Induction |  | 81.8 (8.66)
  Convenience domain Cycle 4 Induction: number analyzed (Participants) | 0 | 11
  Convenience domain Cycle 4 Induction |  | 76.5 (6.26)
  Convenience domain Cycle 5 Induction: number analyzed (Participants) | 0 | 9
  Convenience domain Cycle 5 Induction |  | 79.6 (10.30)
  Convenience domain Cycle 6 Induction: number analyzed (Participants) | 0 | 2
  Convenience domain Cycle 6 Induction |  | 95.8 (5.89)
  Convenience domain Cycle 8 Induction: number analyzed (Participants) | 0 | 43
  Convenience domain Cycle 8 Induction |  | 83.1 (9.18)
  Convenience domain Cycle 2 Treatment: number analyzed (Participants) | 1 | 0
  Convenience domain Cycle 2 Treatment | 75.0 (NA) — The standard deviation could not be calculated from the data of a single participant. |
  Convenience domain Cycle 3 Treatment: number analyzed (Participants) | 30 | 0
  Convenience domain Cycle 3 Treatment | 81.9 (10.28) |
  Convenience domain Cycle 4 Treatment: number analyzed (Participants) | 20 | 0
  Convenience domain Cycle 4 Treatment | 82.1 (12.17) |
  Convenience domain Cycle 5 Treatment: number analyzed (Participants) | 8 | 0
  Convenience domain Cycle 5 Treatment | 83.3 (9.96) |
  Convenience domain Cycle 6 Treatment: number analyzed (Participants) | 13 | 0
  Convenience domain Cycle 6 Treatment | 80.8 (9.85) |
  Convenience domain Cycle 8 Treatment: number analyzed (Participants) | 53 | 0
  Convenience domain Cycle 8 Treatment | 83.8 (11.60) |
  Convenience domain Cycle 2 Maintenance: number analyzed (Participants) | 0 | 33
  Convenience domain Cycle 2 Maintenance |  | 83.6 (8.71)
  Convenience domain Cycle 3 Maintenance: number analyzed (Participants) | 0 | 6
  Convenience domain Cycle 3 Maintenance |  | 87.5 (19.54)
  Convenience domain Cycle 4 Maintenance: number analyzed (Participants) | 0 | 2
  Convenience domain Cycle 4 Maintenance |  | 100.0 (0.00)
  Convenience domain Cycle 5 Maintenance: number analyzed (Participants) | 0 | 8
  Convenience domain Cycle 5 Maintenance |  | 80.2 (12.55)
  Convenience domain Cycle 6 Maintenance: number analyzed (Participants) | 0 | 3
  Convenience domain Cycle 6 Maintenance |  | 83.3 (16.67)
  Convenience domain Cycle 7 Maintenance: number analyzed (Participants) | 0 | 39
  Convenience domain Cycle 7 Maintenance |  | 82.7 (12.59)
  Convenience domain Cycle 8 Maintenance: number analyzed (Participants) | 0 | 4
  Convenience domain Cycle 8 Maintenance |  | 93.8 (12.50)
  Convenience domain Cycle 10 Maintenance: number analyzed (Participants) | 0 | 1
  Convenience domain Cycle 10 Maintenance |  | 91.7 (NA) — The standard deviation could not be calculated from the data of a single participant.
  Convenience domain Cycle 12 Maintenance: number analyzed (Participants) | 0 | 48
  Convenience domain Cycle 12 Maintenance |  | 86.3 (12.69)
  Convenience domain End of Treatment: number analyzed (Participants) | 0 | 3
  Convenience domain End of Treatment |  | 75.0 (16.67)
  Satisfaction domain Cycle 3 Induction: number analyzed (Participants) | 0 | 27
  Satisfaction domain Cycle 3 Induction |  | 89.4 (10.23)
  Satisfaction domain Cycle 4 Induction: number analyzed (Participants) | 0 | 11
  Satisfaction domain Cycle 4 Induction |  | 84.1 (13.80)
  Satisfaction domain Cycle 5 Induction: number analyzed (Participants) | 0 | 9
  Satisfaction domain Cycle 5 Induction |  | 91.7 (8.84)
  Satisfaction domain Cycle 6 Induction: number analyzed (Participants) | 0 | 2
  Satisfaction domain Cycle 6 Induction |  | 93.8 (8.84)
  Satisfaction domain Cycle 8 Induction: number analyzed (Participants) | 0 | 40
  Satisfaction domain Cycle 8 Induction |  | 91.3 (9.47)
  Satisfaction domain Cycle 2 Treatment: number analyzed (Participants) | 1 | 0
  Satisfaction domain Cycle 2 Treatment | 87.5 (NA) — The standard deviation could not be calculated from the data of a single participant. |
  Satisfaction domain Cycle 3 Treatment: number analyzed (Participants) | 30 | 0
  Satisfaction domain Cycle 3 Treatment | 83.3 (11.53) |
  Satisfaction domain Cycle 4 Treatment: number analyzed (Participants) | 20 | 0
  Satisfaction domain Cycle 4 Treatment | 85.6 (13.62) |
  Satisfaction domain Cycle 5 Treatment: number analyzed (Participants) | 9 | 0
  Satisfaction domain Cycle 5 Treatment | 83.3 (8.84) |
  Satisfaction domain Cycle 6 Treatment: number analyzed (Participants) | 13 | 0
  Satisfaction domain Cycle 6 Treatment | 84.6 (14.57) |
  Satisfaction domain Cycle 8 Treatment: number analyzed (Participants) | 54 | 0
  Satisfaction domain Cycle 8 Treatment | 91.2 (12.76) |
  Satisfaction domain Cycle 2 Maintenance: number analyzed (Participants) | 0 | 33
  Satisfaction domain Cycle 2 Maintenance |  | 92.0 (9.28)
  Satisfaction domain Cycle 3 Maintenance: number analyzed (Participants) | 0 | 6
  Satisfaction domain Cycle 3 Maintenance |  | 79.2 (20.41)
  Satisfaction domain Cycle 4 Maintenance: number analyzed (Participants) | 0 | 1
  Satisfaction domain Cycle 4 Maintenance |  | 100.0 (NA) — The standard deviation could not be calculated from the data of a single participant.
  Satisfaction domain Cycle 5 Maintenance: number analyzed (Participants) | 0 | 8
  Satisfaction domain Cycle 5 Maintenance |  | 79.7 (16.28)
  Satisfaction domain Cycle 6 Maintenance: number analyzed (Participants) | 0 | 2
  Satisfaction domain Cycle 6 Maintenance |  | 87.5 (17.68)
  Satisfaction domain Cycle 7 Maintenance: number analyzed (Participants) | 0 | 39
  Satisfaction domain Cycle 7 Maintenance |  | 94.2 (9.00)
  Satisfaction domain Cycle 8 Maintenance: number analyzed (Participants) | 0 | 4
  Satisfaction domain Cycle 8 Maintenance |  | 93.8 (7.22)
  Satisfaction domain Cycle 10 Maintenance: number analyzed (Participants) | 0 | 1
  Satisfaction domain Cycle 10 Maintenance |  | 50.0 (NA) — The standard deviation could not be calculated from the data of a single participant.
  Satisfaction domain Cycle 12 Maintenance: number analyzed (Participants) | 0 | 47
  Satisfaction domain Cycle 12 Maintenance |  | 91.0 (13.21)
  Satisfaction domain End of Treatment: number analyzed (Participants) | 0 | 3
  Satisfaction domain End of Treatment |  | 75.0 (21.65)

ADVERSE EVENTS:
Time Frame: Baseline up to 54 months
Description: Post study start AEs (AEs occurring on the day of or after the first administration of study drug and up to 28 days after the last dose) and is defined as treatment-emergent adverse event (TEAE). All-Cause Mortality is reported for the ITT population
Arm/Group | Diffuse Large B-Cell Lymphoma (DLBCL) | Follicular Lymphoma (FL)
All-Cause Mortality (participants affected / at risk) | 14/72 | 4/86
Serious Adverse Events (participants affected / at risk) | 26/72 | 23/86
Other Adverse Events (participants affected / at risk) | 50/72 | 56/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (DLBCL) (N=72) | Follicular Lymphoma (FL) (N=86)
Neutropenia (Blood and lymphatic system disorders) | 15 | 13
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute Coronary Syndrome (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 0
Klebsiella Infection (Infections and infestations) | 1 | 0
Micrococcus Infection (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil Count Decreased (Investigations) | 5 | 1
White Blood Cell Count Decreased (Investigations) | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Bladder Diverticulum (Renal and urinary disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-Cell Lymphoma (DLBCL) (N=72) | Follicular Lymphoma (FL) (N=86)
Neutropenia (Blood and lymphatic system disorders) | 21 | 20
Anaemia (Blood and lymphatic system disorders) | 11 | 6
Leukopenia (Blood and lymphatic system disorders) | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Pyrexia (General disorders) | 11 | 15
Bronchitis (Infections and infestations) | 1 | 5
Herpes Zoster (Infections and infestations) | 0 | 5
Neutrophil Count Decreased (Investigations) | 9 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Paraesthesia (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 15
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 6
Asthenia (General disorders) | 14 | 3
Influenza Like Illness (General disorders) | 2 | 9
Dysgeusia (Nervous system disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT01889069/SAP_000.pdf
  • Study Protocol (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT01889069/Prot_001.pdf